CLINICAL TRIAL: NCT02269059
Title: A Multiple Dose Study to Evaluate Safety, Pharmacokinetics, and Pharmacodynamics of MK-7680 in Patients With Hepatitis C Infection
Brief Title: Safety and Pharmacokinetics of MK-7680 in Participants With Hepatitis C (MK-7680-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7680-003; 2014-003674-16 (EudraCT Number)
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GT1 Participants (Experimental): Participants take MK-7680 capsules by mouth once daily (QD) for 7 days. The starting dose will be 200 mg and the dose will be adjusted in successive panels of participants based on analysis of results of the previous panel.
  Interventions: Drug: MK-7680
- GT3 Participants (Experimental): Participants take MK-7680 capsules by mouth QD for 7 days. The starting dose will be 200 mg and the dose will be adjusted in successive panels of participants based on analysis of results of the previous panel.
  Interventions: Drug: MK-7680

INTERVENTIONS:
Drug: MK-7680 — MK-7680 10 mg and 100 mg capsules

SUMMARY:
This is a two-part dose-finding trial of MK-7680 in participants with Hepatitis C Virus (HCV) infection of genotype (GT)1 (Part I) and GT3 (Part 2). The primary hypothesis is that daily administration of a safe and well tolerated dose of MK-7680 will produce a decrease in HCV viral load.

DETAILED DESCRIPTION:
Parts 1 and 2 will each consist of 4 panels. In the first panel, a 200 mg dose of MK-7680 will be administered. In each of the following 3 panels, higher or lower doses of MK-7680 will be administered. Each panel will only begin once the safety and tolerability data from the preceding panel have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health except for HCV infection
* Is male or is a female of non-childbearing potential
* Clinical diagnosis of HCV GT1 or GT3 with no evidence of mixed-GT or non-typeable infection

Exclusion Criteria:

* Has a history of clinically significant and not stably controlled endocrine, gastrointestinal, cardiovascular, hematological, hepatic (excepting HCV infection), immunological, renal, respiratory, genitourinary, or major neurological abnormality or disease
* Has a history of cancer
* Has a history of significant multiple and/or severe allergies
* Is positive for hepatitis B or human immunodeficiency virus
* Has had major surgery, donated or lost 1 unit (500 mL) of blood within 4 weeks prior to screening
* Consumes more than 2 alcoholic beverages per day or is currently a regular user of any illicit drug(s) or has a history of alcohol/drug abuse within 12 months prior to screening
* Has chronic hepatitis not caused by HCV (e.g., nonalcoholic steatohepatitis [NASH])
* Has clinical or laboratory evidence of advanced or decompensated liver disease, or evidence of bridging or higher grade fibrosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HCV viral load | Day 1: predose, 2, 4, 8, 12, and 24 hours postdose; Days 3, 4, 5, and 6: predose; and Day 7: predose, 4, 12, 24, and 48 hours postdose
Number of participants experiencing an adverse event (AE) | Up to 21 days
Number of participants discontinuing from study therapy due to AEs | Up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC